CLINICAL TRIAL: NCT06427447
Title: Adjuvant Chemoradiotherapy Versus Chemotherapy for Post-operative Pancreatic Cancer
Brief Title: Adjuvant Chemoradiotherapy Versus Chemotherapy for Pancreatic Cancer (ADJUPANC)
Acronym: ADJUPANC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH hospital
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; adjuvant chemoradiotherapy; adjuvant chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Chemoradiotherapy, Adjuvant; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- adjuvant chemoradiotherapy (Experimental): Chemotherapy: Gemcitabine plus capecitabine Gemcitabine, 1000mg/m2，d1, 8, every 3 weeks as a cycle. Capecitabine, 1650-2000mg/m2，bid, d1-14, every 3 weeks as acycle. A total of 6 cycle should be delivered.
  Chemoradiotherapy: 2-3 weeks after chemotherapy, adjuvant chemoradiotherapy is given. Radiation dose: 50-54Gy (1.8-2.0Gy per fraction). Concurrent capecitabine, 1650mg/m2，bid.
  Interventions: Combination Product: Adjuvant chemoradiotherapy
- adjuvant chemotherapy (Active Comparator): Gemcitabine, 1000mg/m2，d1, 8, every 3 weeks as a cycle. Capecitabine, 1650-2000mg/m2，bid, d1-14, every 3 weeks as acycle. A total of 6 cycle should be delivered.
  Interventions: Drug: Adjuvant chemotherapy

INTERVENTIONS:
Combination Product: Adjuvant chemoradiotherapy — Upfront chemotherapy (gemcitabine plus capecitabine) followed chemoradiotherapy (radiotherapy with concurrent capecitabine)
  Arms: adjuvant chemoradiotherapy
Drug: Adjuvant chemotherapy — Chemotherapy (gemcitabine plus capecitabine)
  Arms: adjuvant chemotherapy

SUMMARY:
In this trial, we aim to compare the outcomes of adjuvant chemoradiotherapy with chemotherapy for patients with resected pancreatic cancer who are at high risk of disease progressions.

DETAILED DESCRIPTION:
Pancreatic cancer is a lethal malignancy with the lowest 5-year overall survival rate of 9% and an increasing incidence. In China, the mortality of pancreatic cancer ranked the sixth among all cancers. Although surgical resection is the only radical treatment, only less than 20% patients could receive upfront surgery at the initial diagnosis. Even though patients have surgery, the incidence of disease progressions, including local progression and metastasis, is about 80-90%. In NCCN guidelines and Chinese guidelines, adjuvant chemotherapy is recommended for post-operative pancreatic cancer, while adjuvant chemoradiotherapy could also be used. However, it has not been clarified that which patients may benefit from adjuvant chemoradiotherapy, and no high-level evidence has shown the advantages of adjuvant chemoradiotherapy over chemotherapy. In meta-analyses, it was demonstrated that patients with lymph nodes metastases, R1 or R2 resection or lymphovascular invasion could achieve longer survival after adjuvant chemoradiotherapy compared with chemotherapy. Therefore, we aim to compare the outcomes of adjuvant chemoradiotherapy with those of chemotherapy in patients with lymph nodes metastases, R1 or R2 resection or lymphovascular invasion after surgical resection of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* Pathologically confirmed pancreatic ductal adenocarcinoma
* Pathologically confirmed lymph node metastasis, R1 or R2 resection or lymphovascular invasion (one of the risk factors)
* No history of cancer treatment after surgical resection
* No disease progression confirmed by imaging examinations
* ECOG 0 to1 point
* No abnormality in blood routine test, liver and kidney function test and coagulation test (White blood cell count ≥4.0×10^9/L, neutrophil count ≥2.0×10^9, hemoglobin level ≥100g/L, platelet count ≥100×10^9/L, ALT and AST level < 2.5 times the upper limit of normal, total bilirubin and creatinine level within the normal, international normalized ratio <2)

Exclusion Criteria:

* History of cancer treatment after surgical resection
* History of other cancers within 5 years
* Disease progression, including local pprogression or metastasis, confirmed by imaging examinations
* ECOG ≥2 points
* Significant abnormality in blood routine test, liver and kidney function test and coagulation test
* Active inflammatory bowel disease
* Gastrointestinal bleeding or perforation within 6 months
* Infections requiring antibiotics
* Heart or respirotory insufficiency
* Pregnant women or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease progression free survival will be determined. | 3 years
  The time from the start of treatment until documentation of any clinical or radiological disease progression or death, whichever occurred first. Progression is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST; version 1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

SECONDARY OUTCOMES:
Overall survival will be determined. | 3 years
  The time from the randomization to death.
Treatment-related adverse events will be determined. | 3 years
  Treatment-related adverse effects are determined by National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Quality of life will be determined. | 3 years
  The analysis of quality of life is based on European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30). All scales and subscales range from 0 to 100. Regarding physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning and global health, higher scores may indicate better outcomes. In the case of fatigue, nausea and vomitting, pain, dyspnea, insomina, appetite loss, constipation, diarrhea and financial difficulties, lower scores may indicate better outcomes. Scales of all items are independent and not combined to compute a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Huojun Zhang, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Huojun Zhang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu X, Liu W, Jiang L, Cao Y, Ye Y, Yu C, Yin X, Zhang H. ADJUPANC protocol: a phase III study of adjuvant chemotherapy versus chemoradiotherapy for pancreatic cancer. Future Oncol. 2025 Aug;21(18):2269-2273. doi: 10.1080/14796694.2025.2522061. Epub 2025 Jun 29. PMID 40583350